CLINICAL TRIAL: NCT03913468
Title: Outcomes of Septic Shock Patients Treated With a Metabolic Resuscitation Bundle Consisting of Intravenous Hydrocortisone, Ascorbic Acid and Thiamine.
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1310; A534285 (Other: UW, Madison); SMPH/MEDICINE/PULMON MED (Other: UW, Madison)
Record Dates: First submitted 2019-02-06; First posted 2019-04-12 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock; Ascorbic Acid Deficiency
Keywords: ascorbic acid; septic shock; severe sepsis
MeSH Terms: conditions — Shock, Septic; Ascorbic Acid Deficiency; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Received Ascorbic Acid IV: Per the medical record, consecutive patients admitted to our institutions ICU with a diagnosis of septic shock within the last 3 years, who were treated within the first 24 hours of admission with the combination of IV ascorbic acid, IV thiamine, and IV hydrocortisone, with a duration of 4 days or until patient leaves the ICU.
  Interventions: Drug: Intravenous Ascorbic Acid
- Control Group: Per the medical record, consecutive patients admitted to our institutions ICU with a diagnosis of septic shock within the last 3 years, who did not receive any treatment with IV ascorbic acid.

INTERVENTIONS:
Drug: Intravenous Ascorbic Acid — 1.5 grams IV ascorbic acid q6h, 50 mg IV hydrocortisone q 6 hours, and 200mg IV thiamine BID administered (as documented in medical record)
  Other Names: Metabolic Resuscitation; HAT therapy
  Groups: Received Ascorbic Acid IV

SUMMARY:
This is a retrospective chart review that will measure the impact on outcomes in septic shock patients who were resuscitated with a novel combination of medicines called iHAT (intravenous hydrocortisone -ascorbic acid-thiamine). Septic shock patients treated with this combination of drugs over the past two years will be compared with similar, concurrent septic shock patients who were not treated with this drug given that adoption of this therapy has been variable.

DETAILED DESCRIPTION:
The condition of septic shock and multi-organ failure directly results from the rapid consumption of ascorbic acid stores in humans suffering an infection (research in septic patients have demonstrated near uniform deficiency/depletion of ascorbic acid on presentation to ICU's).

This rapidly acquired ascorbic acid deficiency leads to shock and multi-organ failure due to the fact that ascorbic acid is required for humans to produce endogenous vasopressors (hormones that regulate blood pressure) as well as to maintain the function and integrity of the endothelium-the endothelium is the largest organ in the body and is critical in regulating blood pressure and preventing fluid leakage into all organs of the body, a pervasive dysfunction which underlies "multi-organ failure". Oral administration of ascorbic acid, even in high doses, has limited bioavailability (transporter mechanisms in the intestines are limited) and does not lead to appreciable correction of the deficiency, neither in the short term, nor in the critically ill.

In contrast, intravenous administration, in high doses, rapidly achieves not only normal levels, but even supranormal levels.This critical need for intravenous supplementation to treat septic shock was first argued for in 2006 by the European Respiratory Society's "Consensus Committee on Intravenous (Parenteral) Vitamin C" a committee comprised of scientists, researchers, and clinicians studying the role ascorbic acid in sepsis/shock models from all over the world. This was followed by two randomized controlled trials in 2014 showing high efficacy of intravenous ascorbic acid in preventing death in septic shock patients. In 2016, a highly publicized historical control trial further demonstrated a large reduction in vasopressor duration, mortality and renal replacement therapy in a cohort of patients after aggressively correcting ascorbic acid deficiency via the intravenous route showing that multi organ failure and death is immediately prevented in almost all patients. More recently, he has published a study demonstrating the synergistic effects of pairing ascorbic acid with hydrocortisone--endothelial barriers are restored to a greater extent than either agent alone.

Lastly, two trials in the past two years have shown that intravenous thiamine, when systematically provided to the critically ill, independently leads to reduced mortality. Thus, HAT therapy appears to be of high utility in preventing death and multi-organ failure in septic shock. Beyond the above mentioned small, single center observational and randomized controlled trials, no other outcome studies have been done in septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitting Provider in the ICU Patient database must be on the Critical Care Service
* Primary diagnosis of sepsis listed in the ICU Patient Database
* Requirement for vasopressors within 24 hours of admission
* If outside transfer, transfer to TLC occurred within 24 hours of initial presentation
* Patient remained on Critical Care service for a minimum of 48 hours
* If treated with iHAT, iHAT started within 36 hours of admission
* No transition to comfort care occurred within the first 24 hours

Exclusion Criteria:

* patients requiring surgical intervention for source control
* patients transitioned to comfort measures only within 24 hours of admission

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU to the medical critical care service with a diagnosis of septic shock
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Duration of Vasopressors | At study conclusion, up to 3 months
  Length of time requiring IV vasopressors

SECONDARY OUTCOMES:
ICU mortality | At study conclusion, up to 3 months
  proportion of patients surviving to ICU discharge
Need for Renal Replacement Therapy | At study conclusion, up to 3 months
  Proportion of patients requiring renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Kory, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No